CLINICAL TRIAL: NCT02023450
Title: Testing of HIV Protease Inhibitors to Suppress Inflammation and Improve Cardio Pulmonary Hemodynamics in Subjects With Pulmonary Arterial Hypertension
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yuan Hong, The Third Xiangya Hospital, The Third Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPI-PAH-0
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Saquinavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- micro/low dose saquinavir and ritonavir (Experimental): To determine if micro dose and low dose SQV+RIT mediates parameters of chronic inflammation in patients with IPAH.
  Interventions: Drug: saquinavir and ritonavir
- standard dose saquinavir and ritonavir (Experimental): To determine if short-term use of SQV+RIT reduces parameters of chronic inflammation and PA pressure of IPAH based on echocardiographic parameters. Safety issue also evaluated at the same time.
  Interventions: Drug: saquinavir and ritonavir

INTERVENTIONS:
Drug: saquinavir and ritonavir — micro and low dose
  Arms: micro/low dose saquinavir and ritonavir
Drug: saquinavir and ritonavir — standard dose
  Arms: standard dose saquinavir and ritonavir

SUMMARY:
Study Rationale:There is recent evidence that HIV protease inhibitors (HIV-PI) can improve pulmonary hemodynamics in experimental models of pulmonary arterial hypertension (PAH). There is also experimental evidence that both TLR4 and high mobility group box 1 (HMGB1) participate in the pathogenesis of experimental pulmonary hypertension. A recent high throughput screen for inhibitors of HMGB1 induced macrophage activation yielded HIV-protease inhibitors (PIs) as potent inhibitors of HMGB1 induced cytokine production. Based on the experimental evidence we propose a trial to determine whether HIV-PIs will alter the pathobiology of PAH.

Study Objectives:The main objective of this study is to determine whether saquinavir and ritonavir (SQV+RIT) which have a well-characterized safety profile in humans will reduce bio markers of inflammation and pulmonary artery pressures in patients with PAH.

Study Hypothesis:We hypothesize that the HIV-PI, SQV+RIT, will reduce circulating parameters of inflammation including HMGB1, IL1-beta, IL-6, IL-8, IL-10, TNF-alpha and CRP. Our end points will be changes in these parameters from baseline over the duration of the study.We hypothesize that treatment with SQV+RIT will reduce pulmonary artery(PA) pressure of patients with PAH as measured by echocardiography.

Study Design:This is a single center open label phase 0 study to evaluate the effect of SQV +RIT in patients with IPAH. Subjects with IPAH(N=20) will be enrolled into a study, which will be divided into 3 cohorts and entail the administration of HIV protease inhibitors in three doses. The first cohort (n=3) will receive a starting dose of SQV 0.3 mg/kg twice daily in combination with RIT 0.03 mg/kg twice daily. If the first dose is well-tolerated, the second cohort (n= 3 ) with IPAH will be given doses of SQV 3 mg/kg and RIT 0.3 mg/kg twice daily. If the second dose is well-tolerated, the last cohort (n= 14 ) with IPAH will be given doses of SQV 15 mg/kg and RIT 1.5 mg/kg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Idiopathic pulmonary arterial hypertension
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study
* Had the diagnosis of PAH confirmed by a cardiac catheterization:Mean pulmonary artery pressure (mPAP) ≥ 25 mm Hg (at rest)，a pulmonary capillary wedge pressure equal or less than 15mmHg, and a normal or reduced cardiac output
* Stable PAH therapy for at least 3 months

Exclusion Criteria:

* Baseline systemic hypotension, defined as MAP less than 50 mmHg
* Required intravenous inotropes within 30 days prior to study participation
* Has uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure >160 mm Hg or sitting diastolic blood pressure >100 mm Hg at screening
* Has a history of portal hypertension or chronic liver disease, including cirrhosis, chronic alcoholism, hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication) defined as moderate to severe hepatic impairment (Child-Pugh Class B-C)
* Has chronic renal insufficiency as defined by serum creatinine >2.5 mg/dL at screening or requires dialysis support
* Has a hemoglobin concentration <9 g/dL at Screening
* History of atrial septostomy
* Repaired or unrepaired congenital heart disease (CHD)
* Pericardial constriction
* Restrictive or congestive cardiomyopathy
* Left ventricular ejection fraction 40% by multiple gated acquisition scan (MUGA), angiography or echocardiography
* Symptomatic coronary disease with demonstrable ischemia
* Other severe acute or chronic medical or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Has a psychiatric, addictive or other disorder that compromises the ability to give informed consent for participating in this study. This includes subjects with a recent history of abusing alcohol or illicit drugs 30 days prior to study screening Day 1 and for the duration of the study
* Poorly controlled asthma defined by active wheezing and/or cough with FEV1 < 70% predicted, responsive to inhaled BD (>15% increase in FEV1 with BD)
* Clinically significant intercurrent illness (including lower respiratory tract infection) or clinically significant surgery within 4 weeks before the administration of study drug
* History of hypersensitivity or idiosyncratic reaction to drugs from multiple drug classes
* Receipt of an investigational product or device, or participation in a drug research study within a period of 15 days (or 5 half lives of the drug, whichever is longer) before the first dose of study drug
* Blood loss or blood donation >550mL within 90 days or plasma donation >500 mL within 14 days before administration of study drug;
* Patients with a QTc interval > 450 msec
* Has diabetes mellitus as defined by symptoms of hyperglycemia and serum fasting plasma glucose level≥7.0mmol/l or casual plasma glucose≥11.1mmol/l at screen
* Has a hyperlipidemia as TC≥6.22 mmol/L, LDL-C ≥4.14 mmol/L or TG ≥2.26 mmol/L
* History of crohn's disease, ulcerative colitis (UC) and etc. Inflammatory bowel disease (IBD)
* Patients who are not willing to take contraceptive measures during the study
* Patients who are taking certain other medication will need to be evaluated for possible exclusion based on the potential for adverse drug interactions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
HMGB1 level | 14 days

SECONDARY OUTCOMES:
TNF、IL-1Β、IL-6、NT-ProBNP and CRP level | 14 days
NYHA/WHO functional class | 14 days
Brog respiration class | 14 days
PA pressure and total right heart function measured by echocardiography | 14 days

OTHER OUTCOMES:
6 minute walk distance | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya hospital, Changsha, Hunan, China

REFERENCES:
- [Derived] Li Y, Li XH, Yu ZX, Cai JJ, Billiar TR, Chen AF, Lv B, Chen ZY, Huang ZJ, Yang GP, Song J, Liu B, Yuan H. HIV protease inhibitors in pulmonary hypertension: rationale and design of a pilot trial in idiopathic pulmonary arterial hypertension. Pulm Circ. 2015 Sep;5(3):538-46. doi: 10.1086/682426. PMID 26401255